CLINICAL TRIAL: NCT07334665
Title: Effects of Posture-Oriented Kinesio Taping on Mobility, Balance, Coordination, and Activities of Daily Living in Patients With Stroke: A Randomized Controlled Trial
Brief Title: Postural Kinesio Taping in Stroke Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, Principal Investigator, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2026-FTR-2
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Hemiplegia; Postural Control
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posture-Oriented Kinesio Taping plus Standard Rehabilitation (Experimental)
  Interventions: Other: Posture-Oriented Kinesio Taping
- Standard Rehabilitation (Active Comparator)
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Other: Posture-Oriented Kinesio Taping — Posture-oriented kinesio taping is applied to trunk and postural muscles to support postural alignment, enhance trunk control, and increase proprioceptive input in patients with stroke. The intervention is delivered as an adjunct to standard neurological rehabilitation and does not replace routine therapy. Kinesio tape is applied by trained clinicians using a standardized posture-focused taping approach, without restricting joint range of motion or limiting functional activities. The taping applications are maintained and renewed at regular intervals throughout the intervention period, with monitoring for skin tolerance and adverse reactions.
  Arms: Posture-Oriented Kinesio Taping plus Standard Rehabilitation
Other: Standard Rehabilitation — Posture-oriented kinesio taping is applied to trunk and postural muscles with the aim of improving postural alignment and trunk control. The taping intervention is administered in addition to a standard neurological rehabilitation program. Applications are performed by trained clinicians using non-elastic-free, hypoallergenic kinesio tape and are renewed at regular intervals during the intervention period. The taping protocol targets postural asymmetry and impaired trunk stability without restricting joint range of motion or limiting functional activities.
  Arms: Standard Rehabilitation

SUMMARY:
Stroke often leads to postural asymmetry and impaired trunk control, which negatively affect mobility, balance, coordination, and activities of daily living. These impairments increase the risk of falls and reduce functional independence during the rehabilitation process.

The purpose of this randomized controlled trial is to investigate the effects of posture-oriented kinesio taping, applied in addition to standard neurological rehabilitation, on functional outcomes in patients with stroke. Participants will be randomly assigned to either an intervention group receiving kinesio taping plus standard rehabilitation or a control group receiving standard rehabilitation alone.

Functional outcomes including trunk control, postural stability, balance, mobility, and activities of daily living will be assessed using validated clinical scales at baseline and after the intervention period. The findings of this study are expected to provide evidence regarding the clinical effectiveness of posture-oriented kinesio taping as a non-invasive and easily applicable adjunct treatment in stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of ischemic or hemorrhagic stroke confirmed clinically and/or radiologically
* In the subacute or chronic phase of stroke (≥1 month post-stroke) and clinically stable
* Presence of postural control and/or trunk control impairment
* Ability to participate in a standard neurological rehabilitation program
* No severe cognitive impairment or communication disorder that would interfere with outcome assessments
* Intact skin at the kinesio taping application sites
* Willingness to participate and provision of written informed consent

Exclusion Criteria:

* Acute stroke phase or clinical instability
* Severe cognitive impairment, aphasia, or insufficient cooperation that would interfere with reliable outcome assessments
* Known allergy or hypersensitivity to kinesio tape
* Active dermatological conditions at taping sites (e.g., open wounds, dermatitis, infection)
* Severe spasticity (Modified Ashworth Scale ≥3)
* Presence of other neurological disorders affecting balance or mobility (e.g., Parkinson's disease, multiple sclerosis)
* Severe orthopedic conditions or cardiopulmonary diseases limiting participation in rehabilitation
* Receipt of posture-oriented kinesio taping within the previous 3 months
* Concurrent participation in another interventional clinical study that could influence study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale (TIS) | Baseline, Week 2, and Week 4
  The Trunk Impairment Scale (TIS) is used to assess trunk control, including static sitting balance, dynamic sitting balance, and trunk coordination in patients with stroke. Higher scores indicate better trunk function.

SECONDARY OUTCOMES:
Postural Assessment Scale for Stroke Patients (PASS) | Baseline, Week 2, and Week 4
  The Postural Assessment Scale for Stroke Patients (PASS) is used to assess postural control and balance during lying, sitting, and standing activities in individuals with stroke. The scale consists of 12 items, with total scores ranging from 0 to 36, where higher scores indicate better postural control and balance performance.
Berg Balance Scale (BBS) | Baseline, Week 2, and Week 4
  The Timed Up and Go Test measures functional mobility and dynamic balance by recording the time required to stand up, walk, turn, and sit down.
10-Meter Walk Test | Baseline, Week 2, and Week 4
  The 10-Meter Walk Test evaluates walking speed as an indicator of functional ambulation.
Functional Independence Measure (FIM) | Baseline, Week 2, and Week 4
  The Functional Independence Measure assesses the level of independence in activities of daily living across motor and cognitive domains.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee YJ, Kim JY, Kim SY, Kim KH. The effects of trunk kinesio taping on balance ability and gait function in stroke patients. J Phys Ther Sci. 2016 Aug;28(8):2385-8. doi: 10.1589/jpts.28.2385. Epub 2016 Aug 31. PMID 27630439